CLINICAL TRIAL: NCT04700566
Title: Safety and Efficacy of Allograft Adipose Matrix Injectable for Glottal Insufficiency
Brief Title: Allograft Adipose Injectable for Vocal Fold Paralysis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Karla O'Dell, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-19-00876
Record Dates: First submitted 2021-01-04; First posted 2021-01-08 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Vocal Fold Palsy
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, interventional clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Injection of Renuva Allograft adipose matrix in vocal fold (Experimental): Injection of Renuva Allograft Adipose matrix in the vocal fold for vocal fold medialization and treatment of glottal insufficiency
  Interventions: Biological: Renuva Allograft Adipose Matrix

INTERVENTIONS:
Biological: Renuva Allograft Adipose Matrix — Injection of Renuva Allograft adipose Matrix in the vocal fold for vocal fold medialization and treatment of glottal insufficiency

SUMMARY:
Renuva is allograft adipose matrix commonly used as a filler in cosmetic procedures.

The investigators are studying this material as an injectable in the vocal fold to treat glottic insufficiency.

Currently, many products can be used as an injectable in the vocal fold to correct glottic insufficiency such as carbomethycellulose, hyaluronic acid, collagen derivatives and calcium hydroxyapatite amongst others. An ideal injectable would not impair the fibroelastic property of the vocal fold tissues and would integrate within the tissue of the vocal fold. Since Renuva has the property of stimulating adipogenesis by using growth factor and collagen, the investigators believe it could represent a good option in terms of safety and efficacy for vocal fold augmentation.

This study will assess the safety and efficacy of Renuva as a vocal fold injectable to treat glottic insufficiency.

DETAILED DESCRIPTION:
Background/Significance:

Vocal cord injection augmentation is commonly used to treat glottal insufficiency. Various materials are used for injection augmentation including autologous fat, hyaluronic acid, collagen, carboxymethylcellulose, and calcium hydroxyapatite. However, all of the current injection choices have individual limitations such as temporary effect, unpredictability due to variable resorption by the body, unfavorable mechanical properties, and challenging handling attributes. Hence, there is a need for a more ideal injection augmentation substance that is biocompatible, nonimmunogenic, able to traverse small gauge needles, easy to use, and facilitates long term or permanent effect when desired.

Intervention:

Unilateral injection augmentation with allograft adipose matrix injectable. Renuva ®, is commonly used as in injectable material in plastic surgery for treatment of small cosmetic irregularities. The injectable stimulates adipogenesis using key matrix proteins including collagen IV, collagen VI, FGF-2, and VEGF. The injectable does not contain any lipids, cellular fragments, or DNA content. In vitro and in vivo demonstrate that the injectable can stimulate adipose tissue generation. Given this important quality, allograft adipose matrix may provide vocal fold bulk for a longer period of time with favorable viscoelastic properties which would make it a desirable agent for vocal fold augmentation.

Objective:

Assess the safety profile and efficacy of allograft adipose matrix for use in injection augmentation Study Design: Single arm prospective clinical trial.

Methods:

50 patients with glottal insufficiency will be enrolled to receive vocal fold augmentation injection using an Allograft adipose matrix, commercially available as Renuva ® over a 24 months recruitment period.

Study endpoints:

Primary study endpoint will be the completion of 12 months of follow up post injection with safety monitoring. Secondary endpoints will include patient reported outcome measures (VHI, VFI, DI and EAT-10), blinded Cape-V voice assessment by experts and laryngeal videostroboscopy blinded assessment with the mVali tool.

Plan for analysis:

The study cohort will be analyzed via descriptive statistics of the primary outcome (safety) via incidence of both minor and major adverse events. Non-parametric statistics (Wilcoxon signed-rank test) will be used for comparisons of patient reported outcome measures and blinded evaluations of voice and videostroboscopy endpoints from post-intervention time points to pre-intervention baseline.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 18 years old

  * Unilateral vocal fold immobility with glottal insufficiency present for at least 2 weeks from onset
  * Willingness to partake in study and follow-up as documented by signed informed consent

Exclusion Criteria:

* History of allergy/hypersensitivity to lidocaine or amide-based anesthetics
* Pregnancy
* Active infection or inflammation in the larynx (presence of acute laryngeal infection caused by bacteria/virus or fungus)
* Comorbid known laryngeal conditions including but not limited to vocal fold scar, vocal tremor, laryngeal dystonia, etc. that would warrant other interventions for optimal treatment
* History of laryngeal surgery
* Life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse recorded in participants after injection | 18 months
  Monitoring of adverse events during the study period for each participant receiving a vocal fold injection with Renuva

SECONDARY OUTCOMES:
Voice outcomes as reported by patient questionnaire | 18 months
  Voice Handicap Index (VHI-10) patient questionnaire at 0, 1, 3, 6, 12, and 18 months
Score on VALI - Voice Vibratory Assessment of laryngeal imaging | 18 months
  Physician assessment of the stroboscopic examination (blinded) using the VALI scaleat day 0, and post injection 1, 3, 6, 12, and 18 months
Dyspnea Index as measured by patient questionnaire | 18 months
  Dyspnea index questionnaired, filled at 0, 1months, 3 months, 6 months, 12 months, 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided